CLINICAL TRIAL: NCT06605898
Title: Optimized Tailored Interventions in Metabolic and Lifestyle Outcomes: Examining the Effects of the Mediterranean-DASH Intervention for Neurodegenerative Delay(MIND) on Cognitive Performance, Metabolic Health and Lifestyle Outcomes Using Advanced Machine Learning Strategies
Brief Title: Optimized Tailored Interventions in Metabolic and Lifestyle Outcomes (OPTIMAL)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Principal Investigator, Naiman Khan, Associate Professor, University of Illinois at Urbana-Champaign
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OPTIMAL
Record Dates: First submitted 2024-09-18; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Change; Diet, Healthy; Metabolic Syndrome, Protection Against
Keywords: Executive function; MIND; Dietary Pattern
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard MIND diet (Experimental): Participants in the active MIND diet group will be asked to consume one ready-to-eat meal per day from Daily Harvest® meal delivery service. This will be a standard treatment arm without prior selection through predictive analytics. The treatment meals will follow MIND diet guidelines and include leafy green vegetables, nuts, legumes, whole grains, berries, and extra virgin olive oil.
  Interventions: Other: MIND Diet
- Predictive Analytics informed MIND Diet (Experimental): Participants in the active MIND diet group informed by predictive analytics will be pre-identified based on the results of a machine learning model that predicts who will most likely benefit from the MIND diet. The participants in this group will be asked to consume one ready-to-eat meal per day from Daily Harvest® meal delivery service. The treatment meals will follow MIND diet guidelines and include leafy green vegetables, nuts, legumes, whole grains, berries, and extra virgin olive oil.
  Interventions: Other: MIND Diet
- Control Diet (Active Comparator): Participants in the control diet group will be asked to consume one ready-to-eat meal per day from Daily Harvest® meal delivery service. The Control group will receive daily meals that are isocaloric with the active/experimental meals but will follow a general diet based on the average American diet and Dietary Guidelines for Americans (i.e., vegetables, fruits, nuts, whole grains, and unsaturated fats).
  Interventions: Other: Control Diet

INTERVENTIONS:
Other: MIND Diet — Daily meals designed to increase adherence to the Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) dietary pattern.
  Arms: Predictive Analytics informed MIND Diet; Standard MIND diet
Other: Control Diet — Daily meals designed to increase fruit, vegetable, and whole grain intake consistent with a healthy American diet.
  Arms: Control Diet

SUMMARY:
The goal of this clinical trial is to learn if increasing adherence to a Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND) diet pattern improves brain and heart health relative to a healthy control diet in middle-aged adults. Our research team will evaluate three different groups: the first group will be chosen using a predictive analytics model that predicts who will benefit most from the MIND diet, the second group will follow the MIND diet without being pre-selected, and the third group will eat a standard healthy diet to serve as a comparison.

The main questions it aims to answer are:

Does the MIND diet improve cognitive performance and heart health relative to a control diet? How does the health impact of the MIND diet in participants pre-identified through predictive analytics compare to those without such pre-selection? Which of the three groups - predictive analytics selected MIND diet group, standard MIND diet group, or healthy control - demonstrate the most significant improvements in cognitive and cardiovascular health over the course of the trial?

Participants will:

Consume one meal that follows the MIND diet or a control meal every day for 3 months. Visit the lab before and after the 3 months of meals for tests. Keep a record of the food they eat during the study.

DETAILED DESCRIPTION:
The purpose of this study is to understand how a healthy diet is related to thinking ability and heart health. Participants will be asked to consume a microwaveable study meal or prepackaged smoothie every day for 12 weeks. These meals will be delivered to participant homes using Daily Harvest meal delivery service. The study meals and smoothies will follow either a dietary pattern thought to improve brain and heart health (MIND), or a control diet, and will include foods commonly found in grocery stores. Participants will not know which diet they are assigned to (active or control). Participants will also be asked to follow simple dietary guidance on a healthy diet in addition to the meals provided. Participants will complete a series of online forms or surveys. Additionally, participants will come to 4 in-person laboratory visits to complete several computer-based tests of memory and attention while wearing an EEG cap. Participants will also be asked to complete an eye test, a heart rate and blood pressure assessment, a bone and body scan called DXA, and a blood draw at the beginning of the study and again at the end of the 12-week diet period.

ELIGIBILITY:
Inclusion Criteria:

* 45-64 years of age
* 20/20 or corrected vision
* No food allergies or intolerances
* Not pregnant, lactating, or have given birth in the past 12 months
* Do not smoke, use tobacco, or abuse drugs
* Absence of liver or gastrointestinal diseases (i.e., primary biliary cirrhosis or gallbladder disease, chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers), hepatitis, HIV, and cancer
* Not currently taking oral hypoglycemic agents, or insulin
* No history of malabsorptive or bariatric surgery
* Cognitively intact with no prior diagnosis of neurological disease (i.e., mild cognitive impairment, Alzheimer's disease, vascular dementia, and/or Asperger's syndrome)
* Able to consume the study meals
* Not enrolled in another dietary, exercise, or medication study during the study.

Exclusion Criteria:

* Non-consent of participant
* Above 64 or below 45 years of age
* Vision not 20/20 or corrected
* Food allergies or intolerances
* Pregnant, lactating, or have given birth in the past 12 months
* Smoke, use tobacco, or abuse drugs
* Prior diagnosis of liver or gastrointestinal disease (i.e., primary biliary cirrhosis or gallbladder disease, chronic constipation, diarrhea, Crohn's disease, celiac disease, ulcerative colitis, irritable bowel syndrome, diverticulosis, stomach or duodenal ulcers), hepatitis, HIV, or cancer
* Currently taking oral hypoglycemic agents or insulin
* History of malabsorptive or bariatric surgery
* Cognitively impaired and/or prior diagnosis of neurological disease (i.e., mild cognitive impairment, Alzheimer's disease, vascular dementia, and/or Asperger's syndrome)
* Unable to consume the study meals
* Concurrent enrollment in another dietary, exercise, or medication study

Ages: 45 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Attentional Accuracy | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in accuracy (%) between groups using a computerized flanker task.
Attentional Reaction Time | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in reaction time (ms) between groups using a computerized flanker task.
Attentional Resource Allocation | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in P3 event related potential amplitude (microvolts) between groups using a computerized flanker task.
Attentional Processing Speed | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in P3 event related potential latency (ms) between groups using a computerized flanker task.
Fasting Blood Glucose | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in fasting blood glucose concentration (mg/dL) between groups.
Fasting Blood Triglycerides | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in fasting blood triglyceride concentration (mg/dL) between groups.
Fasting Blood HDL | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in fasting blood HDL concentration (mg/dL) between groups.
Blood Pressure | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in systolic and diastolic blood pressure (mmHg) between groups
Waist Circumference | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in waist circumference (cm) between groups.

SECONDARY OUTCOMES:
Macular Pigment Optical Density | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in Macular Pigment Optical Density (log units) between groups using a macular densitometer.
Visceral Adipose Tissue | [Time Frame: 12 weeks (Baseline vs Follow-Up)]
  Changes in visceral adipose tissue (g) between groups using Dual X-ray Absorptiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Naiman Khan, PhD, Principal Investigator — University of Illinois Urbana-Champaign
Locations (1):
- University of Illinois at Urbana-Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: No